CLINICAL TRIAL: NCT01849016
Title: N-Acetylcysteine in Patients With Sickle Cell Disease - Reducing the Incidence of Daily Life Pain
Brief Title: N-Acetylcysteine in Patients With Sickle Cell Disease
Acronym: NAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other); Haga Hospital (Other); University Medical Center Groningen (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Fonds NutsOhra (Other); Stichting Janivo (Unknown); CHU Brugmann, Brussels (Other); Erasme University Hospital (Other); Centre Hospitalier Régional de la Citadelle (Other); University Hospital St Luc, Brussels (Other); Centre Hospitalier Universitaire Saint Pierre (Other); Queen Fabiola Children's University Hospital (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, B.J. Biemond, dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NAC trial; 2012-004892-37 (EudraCT Number); 171201003 (Other Grant/Funding Number: ZonMw); NL 41205.018.12 (Other: Central Committee on Research Involving Human Subjects (known by its Dutch initials, CCMO))
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Pain; N-Acetylcysteine; Acetylcysteine; Oxidative stress
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetylcysteine (Experimental): N-Acetylcysteine 600mg 1 oral tablet twice daily during 6 months
  Interventions: Drug: N-Acetylcysteine
- Placebo (Placebo Comparator): Placebo 1 oral tablet twice daily during 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine
  Other Names: Acetylcysteine; Fluimicil; Acetadote
  Arms: N-Acetylcysteine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary aim of this study is to evaluate the effect of the drug N-Acetylcysteine on the frequency of pain in daily life in patients with Sickle Cell Disease (SCD).

Pain is an invalidating hallmark of this disease and has a considerable impact on the Quality of Life of patients and the medical health care system. Oxidative stress is hypothesized to play a central role in its pathophysiology. In pilot studies the administration of N-Acetylcysteine (NAC) resulted in a reduction of oxidative stress. Moreover, administration of NAC seemed to decrease hospitalization for painful crises in a small pilot study in patients with SCD.

This study will be performed as a multicenter, randomized, controlled trial where patients will be treated with either NAC or placebo for a period of 6 months. The investigators expect that NAC can reduce the frequency of pain in patients with SCD, thereby improving their quality of life and participation in society.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years or older
* Sickle cell disease, either homozygous sickle cell disease (HbSS), compound heterozygous sickle cell disease (HbSC), HbSβ0 or HbSβ+ thalassemia
* History of at least 1.0 painful crisis per year in the past 3 years (visit to medical facility is not required)

Exclusion Criteria:

* Chronic blood transfusion or transfusion in the preceding 3 months
* Painful crisis in the last 4 weeks (with respect to the moment of inclusion)
* Pregnancy, breast feeding or the desire to get pregnant in the following 7 months
* Known active gastric/duodenal ulcers
* Hydroxycarbamide (HC) treatment with unstable dose in the last 3 months or started on HC shorter then 6 months prior to study
* Known poor compliance in earlier trials regarding the completion of pain diaries
* Insufficient compliance in run-in period
* Known hypersensitivity to acetylcysteine or one of the other components of the study medication
* Use of pain medication for sickle-cell related pains on more than 15 days per month in the past 6 months ('chronic pain').

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The incidence rate of SCD related pain in daily life per patient year | 6 months
  The incidence of pain in daily life will be expressed as the number of pain days in relation to total follow-up time, and transformed to an event rate per patient year with a corresponding rate ratio and its 95% confidence interval.
  A pain day will be defined as:
  * When the box "Yes, I have experienced pain" is checked in the daily pain diary.
  * Days with hospital admission for painful crisis will be included in the total number of pain days and in the total number of diary observation days, irrespective of pain diary reports on these dates.

SECONDARY OUTCOMES:
The severity of SCD related pain in daily life, using a 0-10 numerical rating scale (NRS) in the study pain diary. | 6 months
  The average intensity of pain indicated on pain days in daily life will be compared between the two groups. The intensity of pain will be calculated as the average pain score over all pain days, using the highest scores indicated per day (either score over night or over day). Hospital days will be excluded from the analysis, as these scores often have not been completed fully during admission and the analysis is targeted at pain in daily life. Pain scores will be considered as continuous data with a normal distribution.
The incidence rate per patient year of painful crises (episodes, based on pain diary observation) | 6 months
  The number of patient-indicated painful crises in relation to total follow-up time will be transformed to an event rate per patient year, with a corresponding rate ratio and it's 95% confidence interval. Also, the average number of crisis days per patient in relation to total follow-up time will be evaluated (including hospital admission days, see below).
  A painful crisis will be defined as either (overlap is possible):
  * When the box "Yes, I was in a crisis" is checked in a daily diary.
  * Missing diary days that are immediately preceded and followed by crisis days or by hospital admission.
  * A visit or admission to a hospital that lasted more than 4 hours for acute sickling-related pain, which was treated with orally or parenterally administered narcotics.
  * An acute chest syndrome
The incidence rate per patient year of days with painful crises (days, based on pain diary observation) | 6 months
  The number of days with patient-indicated painful crises in relation to total follow-up time will be transformed to an event rate per patient year, with a corresponding rate ratio and it's 95% confidence interval.
  A painful crisis will be defined as either (overlap is possible):
  * When the box "Yes, I was in a crisis" is checked in a daily diary.
  * Missing diary days that are immediately preceded and followed by crisis days or by hospital admission.
  * A visit or admission to a hospital that lasted more than 4 hours for acute sickling-related pain, which was treated with orally or parenterally administered narcotics.
  * An acute chest syndrome
The severity of painful crises. This will be defined using a 0-10 numerical rating scale (NRS) in the pain diary. | 6 months
  The average intensity of pain indicated on crisis days in daily life will be compared between the two groups. The intensity of pain will be calculated as the average pain score over all crisis days, using the highest scores indicated per day (either score over night or over day). Hospital days will be excluded from the analysis, as these scores often have not been completed fully during admission and the analysis is targeted at pain in daily life. Pain scores will be considered as continuous data with a normal distribution.
  Painful crisis definition as above.
The incidence rate per patient year of hospital admissions | 6 months
  The number of sickle cell related hospital admissions in relation to total follow-up diary observation time will be transformed to an event rate per patient year, with a corresponding rate ratio and it's 95% confidence interval.
  Admissions will be verified using hospital medical records, if available. Hospital admission will be defined as:
  • Every visit to a hospital that lasted more than 4 hours for acute sickling-related disease, which was treated with orally or parenterally administered narcotics.
The incidence rate per patient year of hospital admission days | 6 months
  The number of sickle cell related hospital admission days in relation to total follow-up diary observation time will be transformed to an event rate per patient year, with a corresponding rate ratio and it's 95% confidence interval.
  Admissions will be verified using hospital medical records, if available. Hospital admission will be defined as:
  • Every visit to a hospital that lasted more than 4 hours for acute sickling-related disease, which was treated with orally or parenterally administered narcotics.
Time in days to first painful crisis (as defined above) | 6 months
  The time in days from randomization to first painful crisis (patient-defined) and hospital admission for painful crisis will be expressed in cumulative event rates, estimated by Kaplan-Meier analysis.
Time in days to first hospital admission for painful crisis (as defined above) | 6 months
  The time in days from randomization to first painful crisis (patient-defined) and hospital admission for painful crisis will be expressed in cumulative event rates, estimated by Kaplan-Meier analysis.
The health-related Quality of Life, as measured by use of validated questionnaires. | 6 months
  In adults this will be assessed with SF36-forms, a short-form health survey that has been proven to be valid and reliable in the black population.46 In children from 12 to 18 years old, we will use the PedsQL questionnaire, often used to assess quality of life in children, also validated in SCD patients
The SCD-related societal costs, assessed by a prospective cost-effectiveness analysis | 6 months
  The societal costs of pain care with the use of NAC, in the intervention group, will be compared to the societal costs of current pain care in the control group. Estimates of unit costs will be based on calculation of real costs of pain care.
  Generated direct medical costs will be recorded in the case record forms and by means of the Medical Cost Questionnaire (see appendix). Indirect costs arising from losses in productivity will be assessed by means of the Productivity Cost Questionnaire (see appendix) and will be calculated by means of the friction cost method.
The tolerability of NAC, defined as the number of participants with adverse events. | 6 months
  This will be assessed via the monthly adverse events reports. The frequency of registered adverse events and/or a serious adverse events will be reported per treatment arm, and compared between the two intervention groups.
The incidence rate per patient year of use of home pain medication (based on pain diary observation). This information will be recorded by subjects in their daily pain diary, including type and dosage of pain medication. | 6 months
  The incidence rate of analgesic usage will be defined as the proportion of pain days with reported analgesic use on the total number of pain days (excluding observation days with no reported pain). This proportion will be transformed to an event rate per patient year, with a corresponding rate ratio and it's 95% confidence interval.
Incidence of SCD complications. | 6 months
  The number of patients with sickle cell related complications (i.e. acute chest syndrome, stroke etc.) will be reported per treatment arm, and compared between the two intervention groups.
  The related incidence of SCD complications;
  * Acute chest syndrome
  * Priapism
  * Hepatic sequestration
  * Splenic sequestration
  * Cerebrovascular accident
  * Leg ulcer
  * Symptomatic avascular osteonecrosis
  These complications will be assessed monthly by using hospital medical records.
The changes in blood markers of oxidative stress, hemolysis, hypercoagulability, inflammation, erythrocyte adhesion and endothelial dysfunction | 6 months
Compliance of study medication; proportion of study medication used based on pill counts. | 6 months
  Compliance of use of study medication will primarily be checked by pill counts (number administered versus number returned). Compliance will be expressed as the proportion of tablets remaining, compared to the number of tablets that should have been taken based on a prescription of 2 tablets per day and the total number of observation days per patient.
Compliance of study medication; N-acetylcysteine plasma concentrations | 6 months
  We additionally aim to evaluate compliance by N-acetylcysteine plasma concentration measurements in blood samples drawn at T0, T3 and T6 in the intervention group, and assess mean change from baseline in the intervention group. This outcome may be used as alternative parameter for patient compliance if pill counts do not suffice.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Biemond, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Karin Fijnvandraat, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (11):
- Belgium (6):
  - CHU Brugmann, Brussels
  - CHU St. Pierre, Brussels
  - Hôpital Erasme, Brussels
  - Hôpital Universitaire Des Enfants Reine Fabiola (HUDERF), Brussels
  - UCL St. Luc, Brussels
  - CHR de la Citadelle, Liège
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
  - Haga Hospital, The Hague
- Guys' & St. Thomas Hospital, London, United Kingdom

REFERENCES:
- [Background] Smith WR, Penberthy LT, Bovbjerg VE, McClish DK, Roberts JD, Dahman B, Aisiku IP, Levenson JL, Roseff SD. Daily assessment of pain in adults with sickle cell disease. Ann Intern Med. 2008 Jan 15;148(2):94-101. doi: 10.7326/0003-4819-148-2-200801150-00004. PMID 18195334
- [Background] Nur E, Brandjes DP, Schnog JJ, Otten HM, Fijnvandraat K, Schalkwijk CG, Biemond BJ; CURAMA Study Group. Plasma levels of advanced glycation end products are associated with haemolysis-related organ complications in sickle cell patients. Br J Haematol. 2010 Oct;151(1):62-9. doi: 10.1111/j.1365-2141.2010.08320.x. Epub 2010 Jul 30. PMID 20678158
- [Background] Nur E, Biemond BJ, Otten HM, Brandjes DP, Schnog JJ; CURAMA Study Group. Oxidative stress in sickle cell disease; pathophysiology and potential implications for disease management. Am J Hematol. 2011 Jun;86(6):484-9. doi: 10.1002/ajh.22012. Epub 2011 May 4. PMID 21544855
- [Background] Nur E, Verwijs M, de Waart DR, Schnog JJ, Otten HM, Brandjes DP, Biemond BJ, Elferink RP; CURAMA Study Group. Increased efflux of oxidized glutathione (GSSG) causes glutathione depletion and potentially diminishes antioxidant defense in sickle erythrocytes. Biochim Biophys Acta. 2011 Nov;1812(11):1412-7. doi: 10.1016/j.bbadis.2011.04.011. Epub 2011 May 3. PMID 21558001
- [Background] Nur E, Brandjes DP, Teerlink T, Otten HM, Oude Elferink RP, Muskiet F, Evers LM, ten Cate H, Biemond BJ, Duits AJ, Schnog JJ; CURAMA study group. N-acetylcysteine reduces oxidative stress in sickle cell patients. Ann Hematol. 2012 Jul;91(7):1097-105. doi: 10.1007/s00277-011-1404-z. Epub 2012 Feb 10. PMID 22318468
- [Background] Pace BS, Shartava A, Pack-Mabien A, Mulekar M, Ardia A, Goodman SR. Effects of N-acetylcysteine on dense cell formation in sickle cell disease. Am J Hematol. 2003 May;73(1):26-32. doi: 10.1002/ajh.10321. PMID 12701116
- [Background] Somjee SS, Warrier RP, Thomson JL, Ory-Ascani J, Hempe JM. Advanced glycation end-products in sickle cell anaemia. Br J Haematol. 2005 Jan;128(1):112-8. doi: 10.1111/j.1365-2141.2004.05274.x. PMID 15606557
- [Background] van Tuijn CF, van Beers EJ, Schnog JJ, Biemond BJ. Pain rate and social circumstances rather than cumulative organ damage determine the quality of life in adults with sickle cell disease. Am J Hematol. 2010 Jul;85(7):532-5. doi: 10.1002/ajh.21731. No abstract available. PMID 20575034
- Available data/document: Statistical Analysis Plan: Version 7.0 - 5/31/2016 — http://www2.hematologie-amc.nl/nac_studie